CLINICAL TRIAL: NCT05371795
Title: Research Study: Tattooing of Skin Landmarks in Radiotherapy: Comparison Between the System Traditional and Comfort Marker 2.0® (COMFORTATTOO)
Brief Title: Comparison on Radiotherapy Permanent Skin Marking With Lancets and an Electric Marking Device
Acronym: COMFORTATTOO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Instituto Portugues de Oncologia, Francisco Gentil, Porto (Other)
Responsible Party: Principal Investigator, André Miranda Pires, Principal Investigator, Instituto Portugues de Oncologia, Francisco Gentil, Porto
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: CONFORTATTOO
Record Dates: First submitted 2022-04-26; First posted 2022-05-12 (Actual); Last update posted 2022-06-10 (Actual); Status verified 2022-06

CONDITIONS: Radiotherapy; Tattooing

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Lancets (Active Comparator)
  Interventions: Device: Lancets
- Comfort Marker 2.0 (Experimental)
  Interventions: Device: Comfort Marker 2.0

INTERVENTIONS:
Device: Comfort Marker 2.0 — The set-up markings are created during the simulation session, after the CT simulation is acquired. For the experimental group, patients' markings are tattooed using an electric marking device developed for set-up marking, the Comfort Marker 2.0® (CM), designed by CIVCO medical solutions, using the 0.2mm deep application depth and the brand-included black pigment. After cleaning the excess ink, if the tattooing was considered unsuccessful, the process was repeated. Markings arrangement followed our departmental protocol. No limit on the maximum number of cutaneous reference points is specified.
  Arms: Comfort Marker 2.0
Device: Lancets — The set-up markings are created during the simulation session, after the CT simulation is acquired. For the control group, patients' markings are tattooed using a 28-gauge disposable lancet and india ink. After cleaning the excess ink, if the tattooing was considered unsuccessful, the process was repeated. Markings arrangement followed our departmental protocol. No limit on the maximum number of cutaneous reference points is specified.
  Arms: Lancets

SUMMARY:
Comparison on radiotherapy skin set-up markings with lancets versus Comfort Marker 2.0®

DETAILED DESCRIPTION:
A Prospective, unicentric, randomized, controlled, parallel, double-blinded, cohort study comparing radiotherapy skin set-up markings with lancets versus electric marking device (Comfort Marker 2.0® by CIVCO®)

ELIGIBILITY:
Inclusion Criteria:

* Age at least 18 years old.
* Patients referred to our department to receive external beam radiation therapy.
* Eastern Cooperative Oncology Group performance status of 0 to 1.
* Estimated fractionating schedule of at least 13 once-daily fractions.
* Written informed consent.

Exclusion Criteria:

* Patients requiring either immobilisation thermoplastic masks (for head or head and shoulders) or vacuum cushion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2021-10-18 (Actual); Primary Completion 2022-03-11 (Actual); Study Completion 2022-09 (Estimated)

PRIMARY OUTCOMES:
Patients' comfort | Day 1
  Comfort is verbally assessed on the 11-point numeric pain scale. As more than one reference point is tattooed, the patients are asked to give an overall score to the procedure.
Effectiveness | up to 7 weeks
  Effectiveness is assessed by the RTT team that delivered the daily fractions. Skin markings are individually evaluated at several periods, specifically at the first fraction, then every 5 fractions, and one last time in the last fraction of RT. These evaluations are scored on a 4-point graded scale (corresponding to bad, reasonable, good, and excellent).

SECONDARY OUTCOMES:
RTTs' satisfaction | Day 1
  The RTT that executed the tattooing is asked to score the ease of the process on a three-point scale (easy, medium, and hard).
Cosmesis | one of the last three days of irradiation
  A photographic assessment is performed. Every set-up marking is individually photographed on one of the last three days of treatment. All photographs are scored by independent observers (both physicians and RTTs) blind to patient identity and treatment allocation, on a five-point scale (corresponding from bad to excellent cosmesis).

OTHER OUTCOMES:
Tattoo fading | 6 months from the end of irradiation
  A photographic assessment is performed. Every set-up marking is individually photographed a. All photographs are scored by indepe6 months after completion of the RT. All photographs are scored by independent observers(both physicians and RTTs) blind to patient identity and treatment allocation, on a five-point scale (corresponding from bad to excellent fading).

CONTACTS AND LOCATIONS:
Locations (1):
- Instituto Português de Oncologia do Porto Francisco Genti, Porto, Portugal

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pires AM, Carvalho L, Santos AC, Vilaca AM, Coelho AR, Oliveira C, Costa C, Fernandes F, Moreira L, Lima J, Vieira R, Ferraz MJ, Silva M, Silva P, Matias R, Zorro S, Costa S, Sarandao S, Barros AF. Radiation Therapy Skin Marking with Lancets Versus Electric Marking Pen (COMFORTATTOO)-6 Months Results on Cosmesis, Fading, and Patients' Satisfaction From a Randomized, Double-Blind Trial. Adv Radiat Oncol. 2023 Nov 5;9(3):101404. doi: 10.1016/j.adro.2023.101404. eCollection 2024 Mar. PMID 38292889

DOCUMENTS (1):
  • Study Protocol and Informed Consent Form (2021-04-10): https://cdn.clinicaltrials.gov/large-docs/95/NCT05371795/Prot_ICF_000.pdf